CLINICAL TRIAL: NCT03878836
Title: Follow-up of Physical, Psychosocial and Cognitive Influences in Persons With Multiple Sclerosis: a Prospective Cohort Study
Brief Title: Follow-up of Persons With Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Serkan Ozakbas, Principal Investigator, Dokuz Eylul University
Other Study IDs: 2959-GOA
Record Dates: First submitted 2019-02-01; First posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Routine assessments — Routine assessments, no specific intervention

SUMMARY:
Multiple sclerosis (MS) is a chronic, progressive and demyelinating disease that affects more than 2.5 million people in the world and is frequently seen in young adults between 20 and 40 years of age, especially in women. Although the exact MS in Turkey is not known, it is estimated as 40/100,000. According to epidemiological studies in recent years, the prevalence and incidence of MS tend to increase. The most common clinical signs and symptoms include loss of sensation in the extremities, partial or total vision loss, acute or subacute motor dysfunction, cognitive impairment, double vision and gait dysfunction.

Currently, MS has no definitive cure. Progressive symptoms related to the disease need to be managed in order to increase and maintain the quality of life of individuals with MS. Pharmacological, physiotherapeutic and psychotherapeutic methods are the most effective effective methods in the management of symptoms. However, the efficacy of these methods has been demonstrated in clinical trials. The outcomes cannot be generalized to the entire MS population because of the inclusion and exclusion criteria that exist in clinical trials. In addition, clinical trials are conducted at a specified time interval (usually a short time interval is selected) and generally, short-term results are provided. In order to better understanding the course of MS, it is of utmost importance that long-term follow-up studies are carried out where as many patients are included and patients are followed from the date of initial diagnosis. The aim of this study is to investigate the change of physical, psychosocial and cognitive characteristics over time and the correlated variables.

The volunteers from MS patients who attend routine control of the MS outpatient clinic of Dokuz Eylül University Hospital will participate in the study. Physical and clinical assessments will be performed by physicians and physiotherapists, and cognitive evaluations will be performed by psychologists with 6-month intervals.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis
* Willingness to participate

Exclusion Criteria:

* Severe cognitive, physical, or psychiatric disability that prevent the assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with multiple sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 118 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Expanded Disability Status Scale | Change from Baseline at 6 Months, 18 Months, 30 Months, 42 Months, and 54 Months
  The Expanded Disability Status Scale is a method of quantifying disability in multiple sclerosis. The scale is based on a neurological examination by a clinician. It has steps from 0 to 10. The higher scores indicate higher neurological disability.

SECONDARY OUTCOMES:
Timed 25-Foot Walk | Change from Baseline at 6 Months, 18 Months, 30 Months, 42 Months, and 54 Months
  The Timed 25-Foot Walk is a quantitative mobility and leg function performance test based on a timed 25-walk. he patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The time is calculated from the initiation of the instruction to start and ends when the patient has reached the 25-foot mark. The task is immediately administered again by having the patient walk back the same distance. Patients may use assistive devices when doing this task. The score is the average of the two completed trials. Higher time represents slower walking speed and more walking impairment.
Timed Up and Go test | Change from Baseline at 6 Months, 18 Months, 30 Months, 42 Months, and 54 Months
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. During the test, the person is expected to wear their regular footwear and use any mobility aids that they would normally require. The time is calculated from the initiation of the instruction to start and ends when the patient has sit down. Higher time represents more static and dynamic balance and mobility impairment.
Single Leg Stance Test | Change from Baseline at 6 Months, 18 Months, 30 Months, 42 Months, and 54 Months
  Single Leg Stance Test measures static balance while standing on a single leg with eyes open and closed. The patient is instructed to remain his/her stability during 60 seconds. The time is recorded while the patient loses his/her stability. The higher time represents better static balance.
6-Minute Walk Test | Change from Baseline at 6 Months, 18 Months, 30 Months, 42 Months, and 54 Months
  The 6-Minute Walk Test is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. The goal is for the individual to walk as far and fast as possible in 6 minutes. The total distance is recorded. Higher distance represents a better submaximal exercise capacity.
12-Item Multiple sclerosis walking scale | Change from Baseline at 6 Months, 18 Months, 30 Months, 42 Months, and 54 Months
  The 12-Item Multiple sclerosis walking scale is a self-assessment scale which measures the impact of multiple sclerosis on walking. It consists of 12 questions with Likert-type choose options concerning the limitations to walking due to multiple sclerosis during the past 2 weeks. Total score ranges 0 from 100. Higher scores indicate more impact of multiple sclerosis on walking.
Modified Fatigue Impact Scale | Change from Baseline at 6 Months, 18 Months, 30 Months, 42 Months, and 54 Months
  The Modified Fatigue Impact Scale provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning. The scale consists of 21 items with a Likert-type choose options. The total score for the scale is the sum of the scores for the 21 items. Individual subscale scores for physical, cognitive, and psychosocial functioning can also be generated by calculating the sum of specific sets of items. The total score ranges from 0 to 84. Higher score indicates higher level of fatigue.
Epworth Sleepiness Scale | Change from Baseline at 6 Months, 18 Months, 30 Months, 42 Months, and 54 Months
  The Epworth Sleepiness Scale is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. The score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the score, the higher that person's average sleep propensity in daily life, or their 'daytime sleepiness'.
Symbol Digit Modalities Test | Change from Baseline at 6 Months, 18 Months, 30 Months, 42 Months, and 54 Months
  The Symbol Digit Modalities Test is used to assess mental processing speed. Higher scores indicate better mental processing speed.
California Verbal Learning Test-II | Change from Baseline at 6 Months, 18 Months, 30 Months, 42 Months, and 54 Months
  The California Verbal Learning Test-II is used to assess verbal memory. Higher scores indicate better verbal memory.
Revised Brief Visuospatial Memory Test | Change from Baseline at 6 Months, 18 Months, 30 Months, 42 Months, and 54 Months
  The Revised Brief Visuospatial Memory Test is used to assess visuospatial memory. Higher scores indicate better visuospatial memory.
Godin Leisure Time Exercise Questionnaire | Change from Baseline at 6 Months, 18 Months, 30 Months, 42 Months, and 54 Months
  The Godin Leisure Time Exercise Questionnaire is a commonly used questionnaire to measure of usual physical activity in persons with multiple sclerosis. It contains three items that measure the frequency of strenuous, moderate, and mild physical activities for periods of more than 15 minutes during one's free time within a typical week. Weekly frequencies of strenuous, moderate and mild physical activity were multiplied by 9, 5 and 3 metabolic equivalents, respectively, and were summed to form a measure of the total leisure physical activity. Scores range from 0 to 864 (hypothetically). Higher scores indicate higher level of physical activity. Participants with 24 units or more are considired as active, 14 - 23 units as Moderately Active, and Less than 14 units as Insufficiently Active/Sedentary.
Multiple Sclerosis International Quality of Life questionnaire | Change from Baseline at 6 Months, 18 Months, 30 Months, 42 Months, and 54 Months
  The Multiple Sclerosis International Quality of Life questionnaire is a disease-specific, self-administered, multidimensional questionnaire, was co-developed and initially validated in 15 countries including Turkey. The questionnaire comprises 31 questions in 9 subscales: activities of daily living, psychological well-being, symptoms, relationships with friends, relationships with family, sentimental and sexual life, coping, rejection, and relationships with healthcare system. All 9 dimensions and the index score were linearly transformed and standardized on a 0-100 scale, where 0 indicates the worst possible level of quality of life and 100 indicates the best level.
Beck Depression Inventory | Change from Baseline at 6 Months, 18 Months, 30 Months, 42 Months, and 54 Months
  The Beck Depression Inventory is a widely used 21-items self-reported measure that assesses the presence and intensity of depressive symptoms reflecting the similar symptoms. Each question has a set of at least four possible answer choices, ranging in intensity. Higher scores indicate higher depressive symptoms. The scores range from 0 to 63.
Nine-Hole Peg Test | Change from Baseline at 6 Months, 18 Months, 30 Months, 42 Months, and 54 Months
  The Nine-Hole Peg Test is used to assess manual dexterity performance. It requires participants to repeatedly place and then remove nine pegs into nine holes, one at a time, as quickly as possible. Two trials for each hand are performed and the score is the average time. Higher scores indicate less manual dexterity performance.
Nordic Musculoskeletal Questionnaire | Change from Baseline at 6 Months, 18 Months, 30 Months, 42 Months, and 54 Months
  The Nordic Musculoskeletal Questionnaire includes 27 items exploring the presence of musculoskeletal symptoms during a 12-month period covering the nine different parts of the body. It also has items pertaining to severity grades, determined according to functional status and the presence of musculoskeletal symptoms during the last 7 days. All answers are given according to a dichotomous 'yes/no' response.
painDETECT Questionnaire | Change from Baseline at 6 Months, 18 Months, 30 Months, 42 Months, and 54 Months
  The painDETECT Questionnaire is used to detect neuropathic pain components.The questionnaire consists of seven questions that address the quality of neuropathic pain symptoms; it is completed by the patient and no physical examination is required. The first five questions ask about the gradation of pain, scored from 0 to 5 (never = 0, hardly noticed = 1, slightly = 2; moderately = 3, strongly = 4, very strongly = 5). Question 6 asks about the pain course pattern, scored from -1 to 2, depending on which pain course pattern diagram is selected. Question 7 asks about radiating pain, answered as yes or no, and scored as 2 or 0 respectively. The final score between -1 and 38, indicates the likelihood of a neuropathic pain component. A score of <=12 indicates that pain is unlikely to have a neuropathic component (< 15%), while a score of >= 19 suggests that pain is likely to have a neuropathic component (> 90%).
International Restless Legs Syndrome Study Group rating scale for restless legs syndrome | Change from Baseline at 6 Months, 18 Months, 30 Months, 42 Months, and 54 Months
  The International Restless Legs Syndrome Study Group rating scale for restless legs syndrome is used to assess severity of the restless legs syndrome symptoms. It consists of 10 items. Higher scores indicate higher severity. The scores range from 0 to 40.

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Ozakbas, MD, Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University Hospital, MS Outpatient Clinic, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided